CLINICAL TRIAL: NCT02648698
Title: A Prospective, Randomized,Controlled Trial on the Effect of Antibiotic Therapy on Endometrial Response in Women With Chronic Endometritis
Brief Title: RCT(Randomized Clinical Trial ) of Antibiotic Therapy in Chronic Endometritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Song Dongmei, Hysteroscopy Center, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FuXingH
Record Dates: First submitted 2015-12-23; First posted 2016-01-07 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Chronic Endometritis
Keywords: chronic endometritis; CD138; antibiotic; conversion rate.
MeSH Terms: interventions — Anti-Bacterial Agents; Levofloxacin; Tinidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic group (Experimental): This group received antibiotic therapy
  Interventions: Drug: Antibiotics
- Control group (No Intervention): This group did not receive antibiotic therapy

INTERVENTIONS:
Drug: Antibiotics — Levofloxacin Tab and Tinidazole Tab are combined in the antibiotic group
  Other Names: Levofloxacin and Tinidazole
  Arms: Antibiotic group

SUMMARY:
120 cases with a diagnosis of chronic endometritis, confirmed by the presence of plasma cells in endometrial biopsy sample identified by immunohistochemical staining using CD138 antibody, have been recruited. The subjects have been randomly divided into two groups, the experimental group have been given antibiotic (Levofloxacin and Tinidazole for 14 days) treatment, the control group did not receive any antibiotic. Initially it was planned for women in the control group to take placebo,but the organization was difficult, so it was changed prior to the start of the study to an open label study. A repeat endometrial biopsy sample have been obtained 2-4 weeks after completion of the antibiotic therapy to assess the response to treatment. The conversion rate will be compared between the two groups

DETAILED DESCRIPTION:
This study will be carried out at the Hysteroscopy centre of the Fuxing Hospital, Capital Medical University ,Beijing, China. A total of 120 women with chronic endometritis who fulfilled the following inclusion criteria will be recruited:

1. CD138 immunohistochemical staining of endometrial specimen showed presence of one or more plasma cells per 10HPF which confirmed chronic endometritis, according to published criteria.
2. women who were pre-menopausal.
3. no evidence of endometrial hyperplasia or malignancy or structural uterine pathology.
4. agreement to have a second endometrial biopsy ~4 weeks after the initial endometrial biopsy.
5. written informed consent obtained

Exclusion Criteria:

1. women who received steroid hormone therapy within one month of recruitment.
2. allergy or suspected allergy to the chosen antibiotic therapy.
3. women who developed any concurrent infection and received any antibiotic therapy during the period of study other than the one prescribed according to the study protocol.

Power calculation: Assuming that the spontaneous CD138 conversion (from positive to negative ) rate is 25% and that the antibiotic therapy results in 60% conversion rate, the total number of subjects required in each arm of the RCT will be 37, accepting a Type I error of 0.05 and a Type II error of 0.1, and assuming a drop-out rate of 20%, 45 subjects will need to be recruited into each arm. Hence, a total of 90 subjects who fulfilled the inclusion criteria will be required.

Recruitment: Women have been recruited form the day case hysteroscopy unit of the Hysteroscopy center, Fuxing Hospital, Beijing, China. The Hysteroscopy center currently carries out ~600 day case hysteroscopy per month. In all cases, endometrial biopsy specimen will be obtained at the time of hysteroscopy for histological evaluation. Since 2013, all endometrial specimens have been routinely examined with the used of CD138 antibody to establish if there is evidence of chronic endometritis, in addition to routine histopathological examination. Previous audit showed that ~15% of subjects had positive staining for CD138 cells.We recruited the initial 132 subjects according to the inclusion and exclusion criteria succesfully from July 2016 to December 2018.

Randomization:Women who had histological confirmation of CE in an endometrial biopsy specimen and who fulfilled the inclusion criteria were randomized into the antibiotic group and control group in a 1:1 ratio using a computer-generated randomization list and sealed opaque envelopes prepared by the first author. The patients were not blinded to the antibiotic treatment. The pathologist who performed the histological evaluation was blinded to the treatment.

Antibiotic therapy: Women who were randomized to the treatment group were given oral Levofloxacin and Tinidazole daily for 14 days.

Women who were randomized to the control group did not receive any antibiotic. Staff Pharmacist dispense medication.

Consent: written informed consent will be obtained

Repeat endometrial biopsy & histological evaluation: The repeat endometrial biopsy will be performed after completion of the the antibiotic therapy. Immunohistochemical study using CD138 antibody will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. CD138 immunohistochemical staining of endometrial specimen showed presence of one or more plasma cells per 10HPF which confirmed chronic endometritis, according to published criteria.
2. women who were pre-menopausal.
3. no evidence of endometrial hyperplasia or malignancy or structural uterine pathology.
4. agreement to have a second endometrial biopsy ~4 weeks after the initial endometrial biopsy.
5. written informed consent obtained

Exclusion Criteria:

1. women who received steroid hormone therapy within one month of recruitment.
2. allergy or suspected allergy to the chosen antibiotic therapy.
3. women who developed any concurrent infection and received any antibiotic therapy during the period of study other than the one prescribed according to the study protocol.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Song, Master, Principal Investigator — FuXing Hospital,Capital Medical University; Enlan Xia, Master, Study Director — FuXing Hospital,Capital Medical University; Tinchiu Li, PhD, Study Chair — FuXing Hospital,Capital Medical University; Xiaoxia Peng, PhD, Study Director — Capital Medical University
Locations (1):
- FuXing Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McQueen DB, Bernardi LA, Stephenson MD. Chronic endometritis in women with recurrent early pregnancy loss and/or fetal demise. Fertil Steril. 2014 Apr;101(4):1026-30. doi: 10.1016/j.fertnstert.2013.12.031. Epub 2014 Jan 23. PMID 24462055
- [Background] Cicinelli E, Matteo M, Tinelli R, Pinto V, Marinaccio M, Indraccolo U, De Ziegler D, Resta L. Chronic endometritis due to common bacteria is prevalent in women with recurrent miscarriage as confirmed by improved pregnancy outcome after antibiotic treatment. Reprod Sci. 2014 May;21(5):640-7. doi: 10.1177/1933719113508817. Epub 2013 Oct 31. PMID 24177713
- [Background] Kitaya K. Prevalence of chronic endometritis in recurrent miscarriages. Fertil Steril. 2011 Mar 1;95(3):1156-8. doi: 10.1016/j.fertnstert.2010.09.061. Epub 2010 Oct 28. PMID 21030015
- [Background] Bayer-Garner IB, Nickell JA, Korourian S. Routine syndecan-1 immunohistochemistry aids in the diagnosis of chronic endometritis. Arch Pathol Lab Med. 2004 Sep;128(9):1000-3. doi: 10.5858/2004-128-1000-RSIAIT. PMID 15335255
- [Background] Kannar V, Lingaiah HK, Sunita V. Evaluation of endometrium for chronic endometritis by using syndecan-1 in abnormal uterine bleeding. J Lab Physicians. 2012 Jul;4(2):69-73. doi: 10.4103/0974-2727.105584. PMID 23440678
- [Background] Kitaya K, Yasuo T. Immunohistochemistrical and clinicopathological characterization of chronic endometritis. Am J Reprod Immunol. 2011 Nov;66(5):410-5. doi: 10.1111/j.1600-0897.2011.01051.x. Epub 2011 Jul 12. PMID 21749546
- [Background] Cicinelli E, Matteo M, Tinelli R, Lepera A, Alfonso R, Indraccolo U, Marrocchella S, Greco P, Resta L. Prevalence of chronic endometritis in repeated unexplained implantation failure and the IVF success rate after antibiotic therapy. Hum Reprod. 2015 Feb;30(2):323-30. doi: 10.1093/humrep/deu292. Epub 2014 Nov 10. PMID 25385744
- [Result] McQueen DB, Perfetto CO, Hazard FK, Lathi RB. Pregnancy outcomes in women with chronic endometritis and recurrent pregnancy loss. Fertil Steril. 2015 Oct;104(4):927-931. doi: 10.1016/j.fertnstert.2015.06.044. Epub 2015 Jul 21. PMID 26207958
- [Derived] Song D, He Y, Wang Y, Liu Z, Xia E, Huang X, Xiao Y, Li TC. Impact of antibiotic therapy on the rate of negative test results for chronic endometritis: a prospective randomized control trial. Fertil Steril. 2021 Jun;115(6):1549-1556. doi: 10.1016/j.fertnstert.2020.12.019. Epub 2021 Feb 3. PMID 33549312
- See also: 2015 — http://www.ncbi.nlm.nih.gov/pubmed/26207958
- See also: 2014 — http://www.ncbi.nlm.nih.gov/pubmed/24462055
- See also: 2013 Oct 31 — http://www.ncbi.nlm.nih.gov/pubmed/24177713
- See also: 2011 Mar — http://www.ncbi.nlm.nih.gov/pubmed/21030015
- See also: 2004 Sep — http://www.ncbi.nlm.nih.gov/pubmed/?term=Routine+syndecan-1+immunohistochemistry+aids+in+the+diagnosis+of+chronic+endometritis
- See also: 2012 Jul — http://www.ncbi.nlm.nih.gov/pubmed/23440678
- See also: 2011 Jul 12 — http://www.ncbi.nlm.nih.gov/pubmed/?term=Immunohistochemistrical+and+clinicopathological+characterization+of+chronic+endometritis
- See also: 2015 Feb — http://www.ncbi.nlm.nih.gov/pubmed/25385744

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 120 subjects were assessed for eligibility. All of the 120 subjects were enrolled and randomized into the antibiotic group and the control group on a 1:1 ratio.
Period: Overall Study
Arm/Group | Antibiotic Group | Control Group
Started | 60 | 60
Completed | 59 | 55
Not Completed | 1 | 5
Not completed — Protocol Violation | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotic Group | Control Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.86 (4.7) | 31.93 (4.8) | 31.89 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 60 | 60 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 59 | 55 | 114
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.91 (3.4) | 22.28 (3.5) | 22.61 (3.4)
Parity [Mean (Standard Deviation); unit: events] | 2.15 (0.9) | 2.15 (0.9) | 2.15 (0.9)
Miscarriage [Mean (Standard Deviation); unit: events] | 1.59 (1.0) | 1.93 (1.0) | 1.75 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: The Conversion Rate of CE (From Positive to Negative)
Description: Subjects in antibiotic group underwent a second-look hysteroscopy and repeat endometrial biopsy for histopathological CD138 immunohistochemical examination 2-4 weeks after completion of antibiotic treatment and in the follicular phase of the following menstrual cycle. Subjects in control group underwent a second-look hysteroscopy and repeat endometrial biopsy for histopathological CD138 immunohistochemical examination ~4 weeks after recruitment in the follicular phase of the following menstrual cycle.
  The biopsies were graded as "negative" for CE if there was less than one plasma cell identified per 10 high-power fields (HPFs) and "positive" when there was one or more plasma cell identified per 10 HPFs.
  To compare the cure rate (From positive to negative) of CE in women who received antibiotic therapy (treatment group) with the spontaneous cure rate in those who did not receive antibiotic therapy (control group),
Time Frame: 1-6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Antibiotic Group: This group received antibiotic therapy
  Women who were randomized to the treatment group were given oral Levofloxacin 500 mg and Tinidazole 1000 mg daily for 14 days.
- Control Group: Women who were randomized to the control group did not receive any antibiotic.
Arm/Group | Antibiotic Group | Control Group
Number analyzed (Participants) | 59 | 55
Percentage of participants | 89.8 [82.2 to 97.5] | 12.7 [3.9 to 21.5]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Antibiotic Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/55
Other Adverse Events (participants affected / at risk) | 0/59 | 0/55

LIMITATIONS AND CAVEATS:
A possible limitation of our study is that patients were not blinded to the antibiotic treatment. A further limitation is the cure rate based on a repeat of test used to make the diagnosis, instead of pregnancy, miscarriage or live birth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT02648698/Prot_SAP_000.pdf